CLINICAL TRIAL: NCT00477815
Title: A Phase I Trial of Zevalin Radioimmunotherapy With High-Dose Melphalan and Stem Cell Transplant for Multiple Myeloma
Brief Title: Rituximab, Yttrium Y 90 Ibritumomab Tiuxetan, Melphalan, and Autologous Peripheral Stem Cell Transplant in Treating Patients With Previously Treated Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000546732; P30CA015083 (NIH); MC048A (Other: Mayo Clinic Cancer Center); 449-05 (Other: Mayo Clinic IRB); NCI-2009-01399 (Registry Identifier: NCI-CTRO); 021-03-ZEV (Other: Biogen IDEC protocol); 106-P148 (Other: Biogen IDEC protocol)
Record Dates: First submitted 2007-05-23; First posted 2007-05-24 (Estimated); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: stage I multiple myeloma; refractory multiple myeloma; stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Rituximab; Melphalan; sargramostim; Granulocyte-Macrophage Colony-Stimulating Factor; ibritumomab tiuxetan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Rituximab + Zevalin (Experimental): Determine the dose level that is both tolerable and achieves the greatest B cell recovery in patients with multiple myeloma.
  Interventions: Biological: rituximab; Drug: melphalan; Biological: Stem Cell; Biological: Sargramostim (GM-CSF); Radiation: 90Y-Zevalin; Biological: 111In Zevalin

INTERVENTIONS:
Biological: rituximab — 375 mg/m2 given as an IV infusion once weekly for four doses (days 1, 8, 15, and 22)
  Other Names: Rituxan, Chimeric Pan-B, C2B8, mouse-human chimeric antibody to CD20 antigen
Drug: melphalan — 100/m2 in 1000 ml 0.9% NaCI IV infusion over 1 hour daily x 2 days.
Biological: Stem Cell — greater than or equal to 2 x 106 CD34+/kg by IV
Biological: Sargramostim (GM-CSF) — 500 mcg by Subcutaneous QD
Radiation: 90Y-Zevalin — Dose escalation scheme. The dose of Zevalin will be based on the calculated radiation to the liver.
  Other Names: Y2B8, 90Y-ibritumomab tiuxetan, IDEC Y2B8
Biological: 111In Zevalin — 5.0 mCi by IV

SUMMARY:
RATIONALE: Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Radiolabeled monoclonal antibodies, such as yttrium Y 90 ibritumomab tiuxetan, can find cancer cells and carry cancer-killing substances to them without harming normal cells. Drugs used in chemotherapy, such as melphalan, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. A peripheral stem cell transplant using stem cells from the patient may be able to replace blood-forming cells that were destroyed by chemotherapy. Giving monoclonal antibody therapy together with chemotherapy and autologous peripheral stem cell transplant may kill more cancer cells.

PURPOSE: This phase I trial is studying the side effects and best dose of yttrium Y 90 ibritumomab tiuxetan when given together with rituximab, melphalan, and autologous peripheral stem cell transplant in treating patients with previously treated multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety of rituximab, yttrium Y 90 ibritumomab tiuxetan, high-dose melphalan, and autologous peripheral blood stem cell transplantation in patients with previously treated multiple myeloma.
* Determine the effect of rituximab and yttrium Y 90 ibritumomab tiuxetan on the clonotypic B-cells at baseline and at B-cell recovery in these patients.

Secondary

* Determine the response rate and progression factors (time to progression, progression-free survival, and duration of response) in patients treated with this regimen.
* Determine the effect of rituximab and yttrium Y 90 ibritumomab tiuxetan on the clonal plasma cells in the blood and marrow prior to high-dose melphalan.

OUTLINE: This is a dose-escalation study of yttrium Y 90 ibritumomab tiuxetan.

Patients receive rituximab IV followed by a dosimetry dose of indium In 111 ibritumomab tiuxetan IV over 10 minutes on day -22. Patients with acceptable biodistribution receive rituximab IV followed by yttrium Y 90 ibritumomab tiuxetan IV over 10 minutes on day -14, high-dose melphalan IV over 1 hour on days -2 and -1, and undergo autologous peripheral blood stem cell transplantation on day 0. Patients also receive sargramostim (GM-CSF) subcutaneously beginning on day 0 and continuing until blood counts recover.

Cohorts of 3-6 patients receive escalating doses of yttrium Y 90 ibritumomab tiuxetan until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Bone marrow, blood, and urine samples are collected at baseline and then periodically during study for biomarker correlative studies.

After completion of study treatment, patients are followed every 3 months for 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of multiple myeloma

  * Previously treated disease
* Candidate for high-dose chemotherapy with melphalan and autologous stem cell transplantation
* No definite evidence of myelodysplasia on pretreatment bone marrow by morphology or by chromosome analysis (e.g., monosomy 7)

  * Chromosome abnormalities from the myeloma clone allowed

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Bilirubin ≤ 2.0 mg/dL
* Alkaline phosphatase ≤ 3 times upper limit of normal (ULN)
* AST ≤ 3 times ULN
* Creatinine ≤ 2 times ULN
* LVEF ≥ 45%
* Corrected pulmonary diffusion capacity ≥ 50%
* No uncontrolled infection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other active malignancy (with the exception of nonmelanoma skin cancer) that requires myelosuppressive chemotherapy or radiation therapy
* No HIV positivity

PRIOR CONCURRENT THERAPY:

* More than 3 weeks since prior myelosuppressive chemotherapy, except cyclophosphamide pulsing for stem cell collection)
* No other concurrent immunotherapy, radiotherapy, chemotherapy or antimyeloma therapy
* Concurrent chronic corticosteroids at doses of prednisone ≤ 20 mg per day (or equivalent) allowed
* Concurrent adjuvant hormonal therapy (e.g., tamoxifen citrate or leuprolide acetate) allowed

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-05-31 (Actual); Primary Completion 2011-07-28 (Actual); Study Completion 2018-05-07 (Actual)

PRIMARY OUTCOMES:
Toxicity as measured by CTCAE v 3.0 | 19 Months
Clonotypic B cells | 19 months

SECONDARY OUTCOMES:
Response (complete response, very good partial response, partial response) | 19 months
Time to progression and duration of response | 5 years
Impact of rituximab and yttrium Y 90 ibritumomab tiuxetan on the clonal plasma cells in the blood and marrow prior to high-dose melphalan | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Angela Dispenzieri, MD, Study Chair — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States